CLINICAL TRIAL: NCT04732936
Title: Feasibility Study of a Temporary Peripheral Nerve Stimulator
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Epineuron Technologies Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EPNR-CIP-001
Record Dates: First submitted 2021-01-19; First posted 2021-02-01 (Actual); Last update posted 2023-07-13 (Actual); Status verified 2023-07

CONDITIONS: Nerve Injury

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Device Usability (Experimental): Device usability and safety will be evaluated.
  Interventions: Device: Temporary Peripheral Nerve Stimulator
- Preliminary Efficacy (Experimental): Preliminary treatment efficacy will be evaluated.
  Interventions: Device: Temporary Peripheral Nerve Stimulator

INTERVENTIONS:
Device: Temporary Peripheral Nerve Stimulator — Temporary Peripheral Nerve Stimulator to deliver 1-hr of electrical stimulation to injured nerves.

SUMMARY:
A novel temporary peripheral nerve stimulator will be evaluated for safety, usability, and preliminary efficacy.

ELIGIBILITY:
Inclusion Criteria:

* Are between 18-65 years old
* Have a Sunderland II-V peripheral nerve injury of the upper extremity
* Are receiving surgery within 14 days of injury

Exclusion Criteria:

* Nerve plexus injuries (e.g. brachial plexus)
* Nerve gap requiring graft/conduit, or extreme joint flexion
* Polyneuropathies
* Cognitive impairment and non-English-speaking
* Uncontrolled diabetes
* Surgical intervention > 14 days of injury
* Co-enrollment in another clinical trial
* Pregnant women

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2021-04-01 (Actual); Primary Completion 2023-06-21 (Actual); Study Completion 2023-06-21 (Actual)

PRIMARY OUTCOMES:
Patient Tolerance to Therapy Questionnaire | Immediately after procedure
Static Two Point Discrimination | 6 months
  Measurement of spatial determination
Semmes-Weinstein Monofilament Test | 6 months
  Measurement of pressure sensitivity
DASH Questionnaire | 6 months
  Validated questionnaire for functionality in upper extremity injury

SECONDARY OUTCOMES:
Safety | 6 months
  As measured by the cumulative incidence of adverse events.
Device Usability Questionnaire | Immediately after procedure

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Coroneos, MD, Principal Investigator — McMaster University
Locations (3):
- Canada (3):
  - Hamilton General Hospital, Hamilton, Ontario
  - McMaster University Medical Centre, Hamilton, Ontario
  - St. Joseph's Healthcare Hamilton, Hamilton, Ontario

REFERENCES:
- [Derived] Coroneos CJ, Levis C, Willand MP, So KJ, Bain JR. Clinical evaluation of a novel disposable neurostimulator used to accelerate regeneration of injured peripheral nerves in the hand. Bioelectron Med. 2025 Apr 25;11(1):9. doi: 10.1186/s42234-025-00171-y. PMID 40275339